CLINICAL TRIAL: NCT03751254
Title: Comparison of Phacoemulsification Platform Stellaris With Standard Infusion and Stellaris Elite With Pressurised Bottle in Myopic Eyes Concerning Deepening of Anterior Chamber as Measured by Intra-operative OCT
Brief Title: Comparison of Stellaris Standard Infusion With Stellaris Elite
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prim. Prof. Dr. Oliver Findl, MBA (Other)
Responsible Party: Sponsor-Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Principal Investigator, Vienna Institute for Research in Ocular Surgery
Organization: Vienna Institute for Research in Ocular Surgery (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Stellaris
Record Dates: First submitted 2018-11-21; First posted 2018-11-23 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Cataract
Keywords: Cataract; Cataract surgery; Phacoemulsification platform
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Myopic patients (Experimental): In myopic patients with axial length over 25.0 mm during surgery of the first eye the Stellaris platform will be used and during surgery of the second eye the Stellaris Elite platform will be used
  Interventions: Device: Stellaris Elite

INTERVENTIONS:
Device: Stellaris Elite — The Stellaris and the Stellaris Elite platform will be used in myopic patients (axial length > 25.0 mm) during cataract surgery

SUMMARY:
Clinical performance of phacoemulsification platform Stellaris Elite with standard irrigation fluid bottles in myopic eyes. Anterior chamber depth and patients comfort will be compared between the two groups.

DETAILED DESCRIPTION:
Today phacoemulsification is the most important and safest procedure to perform cataract surgery. However, there are factors that can increase the risk of complications, one of them is an intraoperative increase of intraocular pressure (IOP) which may cause choroidal haemorrhage, capsular block syndrome, or posterior capsular rupture .

Also, more regularly, alterations of IOP provoke sudden changes of the anterior chamber depth, especially in myopic eyes due to intra-operative inverse irido-capsular block, which may result in pain or discomfort for the patient. The deepening of the chamber also makes the surgical maneuvers more challenging in such eyes.

As prevention of such adverse events, it is important to maintain a more or less constant IOP intraoperatively. To ensure this, the pressure of the irrigation fluid must be adjusted to the outflow of aqueous humor, usually by adapting the height of the irrigation fluid bottle (passive fluidics system). As a variable vacuum is produced at the phaco tip to enable the suction of lens fragments, there often are fluctuations of IOP, therefore the surgeon is required to constantly adjust the height of the irrigation fluid bottle.

A novel method to relieve the surgeon of this often-distracting task is to use all-in-one phacoemulsification systems that are able to monitor vacuum flow rates and then adjust the pressure of the irrigation fluid intraoperatively, also resulting in less fluctuations of IOP (active fluidics system). This should also result in reduced deepening of the anterior chamber and less risk of the adverse events as explained above.

ELIGIBILITY:
Inclusion Criteria:

* Age-related cataract in both eyes
* Scheduled for bilateral cataract surgery
* Myopic patiens with axial eye length >25.0mm
* Age 21 and older
* Written informed consent prior to recruitment

Exclusion Criteria:

* Pregnancy (pregnancy test will be taken pre-operatively in women of reproductive age)
* Preceded ophthalmic surgery
* Any ophthalmic abnormality that could compromise the measurements
* Concurrent participation in another drug or device clinical investigation

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Anterior chamber depth | 12 months
  Anterior chamber depth will be measured using the IOL Master 700. Fluctuations in anterior chamber depth will be compared between the eyes where Stellaris and the contralateral eyes in which the Stellaris Elite platform was used

SECONDARY OUTCOMES:
Patients discomfort | 12 months
  Patients will be asked concerning their discomfort during both cataract surgeries and results will be recorded using an visual analogue scale. In the visual analogue scale 10 means highest discomfort and 1 stands for lowest discomfort.

CONTACTS AND LOCATIONS:
Locations (1):
- Vienna Institute for Research in Ocular Surgery (VIROS), Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided